CLINICAL TRIAL: NCT06464393
Title: The Effect of Opioid-free Anesthesia on Hemodynamic Response and Nociception Level Index During Laryngoscopy and Intubation
Brief Title: Opioid-based Versus Opioid-free Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 548/02-02-2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Anesthesia Intubation; Opioid Use; Analgesic Non-narcotic; Fentanyl
MeSH Terms: interventions — Fentanyl; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine-lidocaine-dexmedetomidine group (Active Comparator): combination of ketamine-lidocaine-dexmedetomidine
  Interventions: Drug: ketamine-lidocaine-dexmedetomidine
- fentanyl group (Active Comparator): fentanyl
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: ketamine-lidocaine-dexmedetomidine — Patients will be administered 0,8 mcg/kg Dexmedetomidine in 100 mL of normal saline within 10 minutes as premedication. Followingly, they will receive 1mL/10 kg of the solution containing ketamine, lidocaine and dexmedetomidine at predefined concentrations just before induction of anesthesia.
  Other Names: KLD group
  Arms: ketamine-lidocaine-dexmedetomidine group
Drug: fentanyl — Patients will be administered 2 mcg/kg fentanyl in 100 mL of normal saline within 10 minutes as premedication. Followingly, they will receive 1mL/10 kg of normal saline solution 0.9% just before induction of anesthesia.
  Other Names: control group
  Arms: fentanyl group

SUMMARY:
The aim of this study will be to investigate the effect of opioid-free induction versus opioid-based induction on hemodynamic response and nociception level index during elective operations

DETAILED DESCRIPTION:
Laryngoscopy and intubation stimuli can cause a sustained sympathetic response manifested as hypertension and tachycardia. Therefore, preadministration of opioid medication aiming at blunting this hemodynamic response is common in everyday anesthetic practice.

Opioid-based anesthesia is associated with side-effects, such as respiratory depression, postoperative nausea and vomiting and occasional induction of tolerance and hyperalgesia.

Research in recent years has focused on the quest for non-opioid-based regimens (opioid-sparing and opioid-free techniques). Most of the relevant studies however focus on the advantages that opioid-free techniques bear on early and late postoperative patient recovery. Literature on the effect of opioid-free techniques especially on laryngoscopy, intubation and subsequent hemodynamic response.

Therefore, the aim of this study will be the comparison of the hemodynamic response to laryngoscopy and intubation between two groups of patients: a group in which opioid medications will be administered before anesthetic induction and a group in which a combination of lidocaine, dexmedetomidine and ketamine will be administered before anesthetic induction.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* American Society of Anesthesiologists (ASA) classification I-II
* Mallampati classification 1, 2 or 3

Exclusion Criteria:

* anticipated difficult airway (Mallampati 4 classification, thyromental distance < 6 cm, mouth opening < 3 cm, neck extension< 80
* atrioventricular block
* bradycardia (heart rate less than 55/min)
* preadministration of beta-blockers
* eligibility for rapid-sequence induction
* chronic use of opioid medications
* known allergy to induction agents
* history of psychiatric disease
* language or communication barriers or lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
change from baseline in systolic arterial pressure after premedication | 30 seconds after premedication
  baseline systolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in systolic arterial pressure immediately after premedication | immediately after intubation
  baseline systolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in systolic arterial pressure 1 minute after intubation | 1 minute after intubation
  baseline systolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in systolic arterial pressure 3 minutes after intubation | 3 minutes after intubation
  baseline systolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in systolic arterial pressure 5 minutes after intubation | 5 minutes after intubation
  baseline systolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in diastolic arterial pressure after premedication | 30 seconds after premedication
  baseline diastolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in diastolic arterial pressure 1 minute after intubation | 1 minute after intubation
  baseline diastolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in diastolic arterial pressure 3 minutes after intubation | 3 minutes after intubation
  baseline diastolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in diastolic arterial pressure 5 minutes after intubation | 5 minutes after intubation
  baseline diastolic arterial pressure will be measured as soon as the patient settles in the operating theatre
change from baseline in heart rate after premedication | 30 seconds after premedication
  baseline heart rate will be measured as soon as the patient settles in the operating theatre
change from baseline in heart rate 1 minute after intubation | 1 minute after intubation
  baseline heart rate will be measured as soon as the patient settles in the operating theatre
change from baseline in heart rate 3 minutes after intubation | 3 minutes after intubation
  baseline heart rate will be measured as soon as the patient settles in the operating theatre
change from baseline in heart rate 5 minutes after intubation | 5 minutes after intubation
  baseline heart rate will be measured as soon as the patient settles in the operating theatre
ST segment change 1 minute post intubation | 1 minute after intubation
  ST segment elevation or depression after intubation
ST segment change 3 minutes post intubation | 3 minutes after intubation
  ST segment elevation or depression after intubation
ST segment change 5 minutes post intubation | 5 minutes after intubation
  ST segment elevation or depression after intubation
duration of nociception level<25 for a 5-minute period after intubation | 5 minutes after intubation
  nociception level (NOL) is a device that measures the status of analgesia intraoperatively. Levels<25 suggest adequate intraoperatively analgesia
time required to achieve a train-of four-ratio of 0 | within 2.5 minutes of neuromuscular blocking agent administration
  the train-of-four (TOF) ratio measures the ratio of the fourth stimulus to the first stimulus of four twitches of neuromuscular stimulation. When this ration reaches the value of 0, the patient is considered ready for intubation

CONTACTS AND LOCATIONS:
Overall Officials: KASSIANI THEODORAKI, PhD, DESA, Principal Investigator — Aretaieion University Hospital, National and Kapodistrian University of Athens, Greece
Locations (1):
- Aretaieion University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shribman AJ, Smith G, Achola KJ. Cardiovascular and catecholamine responses to laryngoscopy with and without tracheal intubation. Br J Anaesth. 1987 Mar;59(3):295-9. doi: 10.1093/bja/59.3.295. PMID 3828177
- [Background] Theodoraki K, Fassoulaki A. Cardiovascular responses to laryngoscopy and tracheal intubation are not accompanied by ST-segment changes. Eur J Anaesthesiol. 2009 Jun;26(6):520-2. doi: 10.1097/EJA.0b013e32831a468d. No abstract available. PMID 19357514
- [Background] Vickovic S, Zdravkovic R, Radovanovic D, Galambos IF, Pap D, Krtinic D, Stanisavljevic S, Preveden M, Videnovic N, Videnovic J. Effect of different doses of remifentanil on the cardiovascular response after endotracheal intubation: a randomized double-blind study. Eur Rev Med Pharmacol Sci. 2023 Jan;27(2):653-658. doi: 10.26355/eurrev_202301_31067. PMID 36734737
- [Background] Feenstra ML, Jansen S, Eshuis WJ, van Berge Henegouwen MI, Hollmann MW, Hermanides J. Opioid-free anesthesia: A systematic review and meta-analysis. J Clin Anesth. 2023 Nov;90:111215. doi: 10.1016/j.jclinane.2023.111215. Epub 2023 Jul 27. PMID 37515877
- [Background] Patel J, Snyder K, Brooks AK. Perioperative pain optimization in the age of the opioid epidemic. Curr Opin Anaesthesiol. 2024 Jun 1;37(3):279-284. doi: 10.1097/ACO.0000000000001370. Epub 2024 Mar 12. PMID 38573179